CLINICAL TRIAL: NCT04351009
Title: Intra-operative Sentinel Lymph Node Mapping Using Indocyanine Green Dye Near-infrared Fluorescence Imaging in Colon Cancer: Prospective Single Center Study
Brief Title: Sentinel Lymph Node Mapping and Analysis in Colon Cancer Using Indocyanine Green Dye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICG001
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Colon Cancer
Keywords: Sentinel lymph node; Indocyanine green
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Sentinel lymph node mapping: 25 mg of Indocyanine green dye diluted in 1 ml of 20% Albumin solution and 9 ml of 0.9% Normal saline solution will be used. Injections (0.5-1 ml) will be given in the submucosa or subserosa at 2-4 points around the tumor proximally and distally. Lymphatic flow will be followed after injection in real time with Near-infrared fluorescence imaging scope until sentinel lymph nodes will be identified.
Masking Description: The pathologist involved in routine histological assessment of the resected lymph nodes including lymph nodes in the gross specimen and sentinel lymph nodes will be blinded to the identity of the sentinel lymph nodes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine green sentinel lymph node mapping (Experimental): Indocyanine green dye is injected in the submucosa or subserosa around the tumor to identify sentinel lymph nodes intra-operatively with near infrared fluorescence imaging.
  Interventions: Procedure: sentinel lymph node mapping

INTERVENTIONS:
Procedure: sentinel lymph node mapping — Through on-table colonoscopy indocyanine green solution will be injected in the submucosa at 2-4 points around the tumor for laparoscopic surgeries. Dye will be injected in the subserosa at 2-4 points for open surgeries. Lymphatic flow from the tumor will be mapped in real time with near-infrared fluorescence imaging scope and sentinel lymph nodes will be identified.

SUMMARY:
Approximately 20-30 % of colon cancer patients who have no metastasis in lymph nodes after definitive colectomy have recurrence with distant metastasis. These recurrences could be due to missed occult tumor cells or micrometastasis. Detailed examination of all lymph nodes is expensive and time consuming. Sentinel lymph node mapping using Indocyanine green dye helps in identifying the lymph nodes which are most likely to harbour metastasis. These sentinel lymph nodes can be subsequently subjected to detailed pathologic examination and immunohistochemistry which increases the likelihood of identifying micrometastasis and occult tumor cells. Patients found to harbour such metastasis can be treated with additional chemotherapy after surgery. The aim of the study is to examine the feasibility of sentinel lymph node mapping using Indocyanine green dye in colon cancer and evaluate the upstaging rate in post-operative colon cancer patients who don't have metastatic lymph nodes on routine histopathology.

DETAILED DESCRIPTION:
All patients of colon cancer fulfilling the inclusion criteria and excluding the patients according to the exclusion criteria will undergo standard laparoscopic/open colectomy.

Indocyanine green dye is injected around the tumor in subserosal location for open surgeries and submucosally after on-table colonoscopy for laparoscopic surgeries and followed with near-infrared scope. Patients will undergo intra-operative on-table colonoscopy after induction of anesthesia. All sentinel nodes will be marked with clips/sutures for identification by the pathologist post-operatively. Any aberrant lymph nodes identified outside the planned resection margins will be excised, marked with the position of excision and sent separately from the gross specimen. After this the surgeon will proceed with the surgery including vascular ligation and resection of mesocolon.

After surgery, all the lymph nodes identified in the specimen including the tagged sentinel lymph nodes will be examined using standard Hematoxylin and eosin staining. If all the lymph nodes are negative for metastasis, the sentinel lymph nodes will undergo additional stepwise sections and immunohistochemistry for pancytokeratin.

ELIGIBILITY:
Inclusion criteria:

Age 18 years or older Biopsy proven colon cancer Scheduled for laparoscopic/open colectomy

Exclusion criteria:

Prior colorectal surgery Gross lymph node invasion on pre-operative imaging or intraoperative staging Advanced disease (T4 disease or metastasis) on preoperative imaging or intraoperative staging Allergy to iodide containing compounds, human albumin or Indocyanine green dye History of hyperthyroidism or thyroid adenoma Palliative surgery Advanced hepatic failure Advanced renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Detection rate | 2 years
  Proportion of the number of successful sentinel lymph node procedures out of all executed sentinel lymph node procedures.
Upstaging rate | 2 years
  Sentinel lymph nodes in patients are pathologically node negative on routine evaluation with undergo detailed evaluation using serial sections and immunohistochemistry to identify micrometastasis and occult tumor cells. The proportion of node negative patients who are upstaged will be calculated.

SECONDARY OUTCOMES:
Accuracy | 2 years
  No of patients with successful sentinel lymph node mapping - False negatives/ No of patients with successful sentinel lymph node mapping.
Negative predictive value | 2 years
  number of patients in whom a negative sentinel lymph node correctly predicted the lymph node status of the total lymph node yield.
Aberrant lymph node drainage | 2 years
  proportion of sentinel lymph nodes identified outside planned resection margins and their tumor bearing status .

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev M Patil, MS, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No